CLINICAL TRIAL: NCT06664463
Title: Reviving Hope: Rehabilitation of Traumatic Brain Injury: Nursing Approaches for Arousal Enhancement
Brief Title: Impact of Sensory Stimulation Techniques on Consciousness Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Elsayed Zaky, Principle investiagtor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Arousal Recovery
Record Dates: First submitted 2024-10-22; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Trumatic Brain Injury
Keywords: stimulation techniques; Recovery; nursing role

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): * This study group will undergo an Arousal Enhancement Protocol, designed to increase physiological and psychological arousal in unconscious patients. Participants will be exposed to controlled stimuli, such as visual or auditory tasks, while their responses are monitored using devices to measure heart rate temparature, blood pressure and respiratory rate.
  * No drug interventions are involved in this protocol, with a focus on non-invasive sensory stimulation techniques. The goal is to understand how enhanced arousal affects physiological responses and promotes recovery. Participation is conducted with a focus on safety and strict adherence to ethical guidelines
  Interventions: Other: Arousal enhancment protocol
- Control Group (Placebo Comparator): group that will recieve routine hospital care
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Arousal enhancment protocol — Auditory stimulation: Playing familiar music or personalized playlists tailored to the patient's preferences evokes emotional responses and promotes arousal.
  Olfactory stimulation: Using essential oils or fragrances associated with calming or invigorating properties fosters emotional connections and evokes nostalgia through scents linked to positive memories.
  Visual stimulation: Displaying photographs of family members or significant events provides comforting visual stimulation and stimulates visual awareness.
  Tactile stimulation: Gentle touch or therapeutic massage engages the patient through tactile input, promoting physiological and emotional responses.
  Besid thsi protocl also the will recivce routine care throughout study period The control group in this study will receive routine hospital care. This care includes standard medical evaluations, monitoring of vital signs, neurological assessments, and any necessary imaging (such as CT or MRI scans). Patients will also receive s
  Arms: Study group
Other: Routine Care — The control group in this study will receive routine hospital care. This care includes standard medical evaluations, monitoring of vital signs, neurological assessments, and any necessary imaging (such as CT or MRI scans). Patients will also receive supportive care, including pain management, hydration, and nutrition, as well as physical, occupational, or speech therapy as needed based on their recovery progress
  Arms: Control Group

SUMMARY:
Traumatic brain injury is a leading cause of long-term disability, necessitating innovative rehabilitation methods. This study evaluates the effectiveness of integrating nursing techniques with arousal enhancement protocol to promote neurological recovery in traumatic brain injury patients.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a significant global health concern, often leading to long-term disabilities that severely impact daily functioning and quality of life. Patients with traumatic brain injury frequently experience altered states of consciousness, complicating rehabilitation efforts and necessitating innovative approaches to care. Traditional rehabilitation strategies often emphasize physical recovery and may overlook the potential of sensory stimulation in enhancing cognitive function and arousal.

The arousal enhancement protocol represents a promising framework that integrates sensory modalities to actively engage patients in their rehabilitation. By focusing on personalized, nurse-led interventions, this protocol aims to foster greater patient involvement and optimize recovery outcomes. However, there is a pressing need for systematic evaluation of these approaches to better understand their efficacy and long-term impact on patient recovery.

Background Traumatic brain injury is a leading cause of long-term disability, significantly impacting patients' quality of life and daily functioning. Despite advancements in medical care, many individuals with TBI remain in a state of impaired consciousness, complicating their rehabilitation and recovery. Current rehabilitation strategies often lack the integration of nursing approaches specifically aimed at enhancing arousal and responsiveness in these patients. This gap highlights the need for innovative nursing interventions that incorporate structured sensory stimulation techniques to promote neurological recovery. The effectiveness of such approaches in improving arousal levels and cognitive function in patients with traumatic brain injury has not been thoroughly evaluated, necessitating research that explores the role of nursing in implementing arousal enhancement protocols. This study aims to address this issue by assessing the impact of nursing-led sensory stimulation interventions on the recovery outcomes of patients with traumatic brain injury, thereby reinforcing the critical role of nursing in optimizing rehabilitation strategies for this vulnerable population.

The arousal enhancement protocol refers to a series of structured interventions aimed at promoting the recovery of patients with traumatic brain injury who have reduced levels of consciousness. The protocol includes sensory, cognitive, and physical stimulation techniques administered to engage the patient's senses and stimulate brain activity. In this study, techniques such as auditory, visual, olfactory, and tactile stimulation were utilized to increase the responsiveness of patients with traumatic brain injury, ultimately enhancing their cognitive and neurological recovery.

The arousal enhancement protocol encompasses a diverse range of interventions aimed at awakening and engaging individuals who have lapsed into a coma following a traumatic brain injury. These techniques are designed to promote arousal, sensory awareness, and cognitive responsiveness in patients with impaired consciousness. Common approaches include sensory stimulation, such as auditory, visual, olfactory, and tactile stimuli, which were applied in this study in a structured and systematic manner to evoke responses and increase arousal levels.

At the heart of this intervention lies the pivotal role of nursing professionals, whose expertise, compassion, and dedication are instrumental in driving the success of the program. Nursing involvement in the arousal enhancement protocol for traumatic brain injury rehabilitation represents a fusion of clinical skill, therapeutic insight, and patient-centered care. The application of the arousal enhancement protocol in traumatic brain injury rehabilitation represents a pioneering frontier in nursing practice. Throughout the implementation of the arousal enhancement protocol, nurses play a central role in the delivery of sensory stimuli tailored to each patient's unique preferences and responses. From gentle touch and therapeutic massage to auditory stimulation and olfactory cues, nurses harness a diverse array of modalities to engage patients in the rehabilitation process. Their adeptness in therapeutic communication fosters a nurturing and supportive environment conducive to patient participation and progress.

Moreover, nurses play a critical role in the rehabilitation process. They meticulously document changes in arousal levels, vital signs, and behavioral indicators, ensuring that these observations guide timely adjustments to the stimulation protocol. This data-driven approach optimizes the effectiveness of the intervention while mitigating potential risks. Additionally, nurses implement targeted rehabilitation techniques, such as sensory re-education and motor relearning exercises, tailored to the patient's specific needs. They collaborate closely with interdisciplinary team members, including physicians, therapists, and caregivers, to ensure seamless coordination of care and holistic support for patients and their families, thus facilitating a comprehensive and integrated rehabilitation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years.
* Suffering from traumatic brain injury.
* With stable vital signs within normal ranges.
* Having a Glasgow Coma Scale (GCS) score of 9 or more.
* Admitted to the inpatient neurology department.

Exclusion Criteria:

* Individuals with a GCS score of less than 9.
* Individuals with deafness, blindness, aphasia, hemiplegia, or quadriplegia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Glasgo Coma Scale | 2 weeks
  * The Glasgow Coma Scale (GCS) is a clinical tool used to assess a person's level of consciousness following a brain injury. It evaluates three key areas: eye opening, verbal response, and motor response.
  * Scoring : The GCS assigns a score in each category, with a total score ranging from 3 to 15, where:
  Severe brain injury: 3-8 Moderate brain injury: 9-12 Mild brain injury: 13-15

SECONDARY OUTCOMES:
Western Neuro Sensory Stimulation Profile | 2 weeks
  * The Western Neuro Sensory Stimulation Profile (WNSSP) is a standardized assessment tool used to evaluate the sensory and cognitive responsiveness of patients with severe brain injuries, including traumatic brain injury (TBI). It measures outcomes related to sensory awareness, arousal, and cognitive function by assessing patient responses to various sensory stimuli, such as auditory, visual, tactile, and olfactory cues. The WNSSP provides valuable insights into a patient's level of consciousness and recovery progress, helping clinicians tailor rehabilitation strategies and monitor improvements in responsiveness over time.
  * Scoring: The WNSSP has a scoring range from 0 to 113, where higher scores indicate better outcomes. Specifically, higher scores reflect greater levels of sensory awareness and cognitive responsiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Faculy of Nursing Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seo NJ, Ramakrishnan V, Woodbury ML, Bonilha L, Finetto C, Schranz C, Scronce G, Coupland K, Blaschke J, Baker A, Howard K, Meinzer C, Velozo CA, Adams RJ. Concomitant sensory stimulation during therapy to enhance hand functional recovery post stroke. Trials. 2022 Apr 5;23(1):262. doi: 10.1186/s13063-022-06241-9. PMID 35382902
- See also: Related Info — https://journals.lww.com/jinm/fulltext/2024/06020/impact_of_auditory_stimulation_nursing_protocol_on.7.aspx?context=latestarticles